CLINICAL TRIAL: NCT00390403
Title: A Phase I, Open Label Study of AT-101 Plus Radiotherapy and Temozolomide and of AT-101 Plus Adjuvant Temozolomide for Patients With Newly-Diagnosed Glioblastoma Multiforme
Brief Title: Gossypol (AT-101) and Temozolomide With or Without Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NABTT-0602 CDR0000507451; U01CA062475 (NIH); NABTT-0602
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult gliosarcoma; adult giant cell glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Temozolomide; Gene Expression Profiling; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: R-(-)-gossypol acetic acid
Drug: temozolomide
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: protein expression analysis
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gossypol and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Gossypol may help temozolomide work better by making tumor cells more sensitive to the drug. Gossypol may also make tumor cells more sensitive to radiation therapy. Giving gossypol and temozolomide together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of gossypol when given together with temozolomide with or without radiation therapy in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of gossypol (AT-101) when administered with radiotherapy (RT) and concurrent temozolomide (TMZ) in patients with newly diagnosed glioblastoma multiforme.
* Determine the MTD of gossypol when administered with adjuvant TMZ after standard RT and concurrent TMZ in these patients.

Secondary

* Assess the toxicity of these treatment regimens.
* Assess and describe the pharmacokinetics of gossypol.
* Determine, preliminarily, the therapeutic activities of these regimens.
* Determine the relationship between these regimens and cellular and molecular features identified in tumor biopsy specimens.

OUTLINE: This is a multicenter, open-label, nonrandomized, dose-escalation study of gossypol. Patients are assigned to 1 of 2 treatment groups. Patients who participate in group I are NOT eligible for group II.

* Group I: Patients receive oral gossypol and undergo radiotherapy once daily 5 days a week for up to 6 weeks. Patients also receive oral temozolomide once daily for up to 6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
* Group II: Patients receive oral temozolomide on days 1-5 and oral gossypol once daily on days 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-10 patients per treatment group receive escalating doses of gossypol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 or 3 of 10 patients experience dose-limiting toxicity.

Patients undergo blood collection periodically for pharmacokinetic studies. Tumor tissue samples are examined for biomarkers including, but not limited to, Bcl-2 family protein expression (e.g., Bcl-2, Bcl-xL, MCl-1, Bax, Bak, and BH3 domain), MGMT gene methylation status, and gene expression array.

After completion of study treatment, patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial grade IV astrocytoma (glioblastoma multiforme)
* Meets 1 of the following criteria:

  * Completed surgery within the past 6 weeks (group I)
  * Received radiotherapy and concomitant temozolomide at least 4 weeks but no more than 7 weeks prior to start of study treatment (group II)
* Must be on a stable corticosteroid regimen (no increase for 5 days)

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Hemoglobin ≥ 10 g/dL
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤1.5 mg/dL
* Bilirubin ≤ 1.5 mg/dL
* ALT and AST ≤ 2.5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after completion of study treatment
* Mini Mental State Exam score ≥ 15
* Must be able to swallow and retain oral medication
* No serious concurrent infection or medical illness that would preclude study participation
* No other malignancy within the past 5 years, except for curatively treated carcinoma in situ or basal cell carcinoma of the skin
* No sensory neuropathy ≥ grade 2
* No allergies to gossypol
* No symptomatic hypercalcemia or hypercalcemia > grade 2
* No gastrointestinal disease including any of the following:

  * Malabsorption syndrome
  * Disease significantly affecting gastrointestinal function
  * Ulcerative colitis
  * Inflammatory bowel disease
  * Partial or complete small bowel obstruction

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from the immediate postoperative period
* No prior radiotherapy, chemotherapy, immunotherapy, therapy with biologic agents (including immunotoxins, immunoconjugates, antisense agents, peptide-receptor antagonists, interferons, interleukins, tumor-infiltrating lymphocyte therapy, lymphokine-activated killer cells or gene therapy), or hormonal therapy for this brain tumor (group I)

  * Prior glucocorticoid therapy allowed
* No prior polifeprosan 20 with carmustine implant (Gliadel wafers) (group I)
* No prior gossypol
* No prior radiosurgery or brachytherapy
* No prior resection of the stomach or small intestine
* No other concurrent anticancer therapy (i.e., chemotherapeutics or investigational agents)
* No concurrent cytochrome p450 enzyme-inducing anticonvulsant drugs
* No concurrent prophylactic filgrastim (G-CSF)
* No concurrent iron supplements

  * Nutritional supplements containing iron allowed
* No concurrent intensity-modulated radiotherapy
* No concurrent electron, particle, implant, or stereotactic radiosurgery boost

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose

SECONDARY OUTCOMES:
Toxicity
Pharmacokinetic profile of gossypol
Therapeutic activity
Cellular and molecular outcomes (intratumoral expression levels of biomarkers, including Bcl-2 family protein expression [e.g., Bcl-2, Bcl-xL, MCl-1, Bax, Bak, BH3 domain], MGMT gene methylation status, and gene expression array)

CONTACTS AND LOCATIONS:
Overall Officials: John Fiveash, MD, Study Chair — University of Alabama at Birmingham
Locations (8):
- United States (8):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania